CLINICAL TRIAL: NCT05919290
Title: HN QUEST- Evaluation of Online MRgRT and Repeat Functional Imaging in Patients Undergoing Curative (CT)RT for HN Malignancy
Brief Title: HN-QUEST: A Study of Head and Neck Imaging Biomarkers
Acronym: HN-Quest
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-5864
Record Dates: First submitted 2023-01-08; First posted 2023-06-26 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HNSCC patients (Other): Up to 100 HNSCC patients receiving CT-based radiation therapy will receive up to weekly non-contrast MRI scans during treatment.
  Interventions: Other: MRI
- Healthy volunteers and HNSCC patients (Other): Cohort A - Up to 20 healthy volunteers will undergo non-contrast MRI at two time points.
  Cohort B - Up to 53 patients planned to receive curative (chemo) radiotherapy for HNSCC will undergo two baseline MRI scans, one MRI in week 2 and week 4, and final MRI scan 6-8 weeks after completion of treatment.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Non-invasive imaging technique that is used to take pictures of organs within the body.

SUMMARY:
This is a multi arm, single center, investigator initiated study to investigate online adaptive radiotherapy and biomarker development in patients with newly diagnosed HNSCC (Head and Neck Squamous Cell Carcinoma) receiving curative therapy.

The study will consist of two prospective arms. In Arm 1 up to 100 HNSCC patients receiving (CT)RT (computed tomography-based radiation therapy) will receive up to weekly non-contrast MRI (magnetic resonance imaging) scans during treatment. Arm 2 consists of two cohorts. In cohort A up to 20 healthy volunteers will undergo non-contrast MRI at two time points. In cohort B up to 53 patients planned to receive curative (chemo) radiotherapy for HNSCC will undergo two baseline MRI scans, one MRI in week 2 and week 4, and final MRI scan 6-8 weeks after completion of treatment.

DETAILED DESCRIPTION:
The purpose of this study is to develop and investigate novel and established MR (magnetic resonance) imaging sequences as predictive and prognostic radiotherapy biomarkers. Radiotherapy is a fundamental treatment modality for Head and Neck Squamous Cell Carcinoma (HNSCC) with a majority of patients receiving radiation as part of their care pathway. Although treatment is effective, there remains a risk of failure particularly in those presenting with locally advanced disease. In addition, significant proportion of patients receiving radiotherapy will suffer long-term side effects related to their treatment. The addition of concurrent chemotherapy improves the efficacy of radiotherapy, but at the cost of increased treatment related toxicity. The treatment related toxicity and risk of treatment failure means there is a compelling clinical need to personalize therapy based on a patient's early response to radiotherapy.

ELIGIBILITY:
Inclusion Criteria for Cancer Patients:

* Age >/= 18 years
* Histologically proven Head and Neck Squamous Cell carcinoma
* Primary or nodal disease > 3cm for biomarker imaging
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Planned for curative surgery or (chemo)radiotherapy
* Willingness to undergo repeat MRI
* Able to receive and understand verbal and written information regarding study and able to give written informed consent
* Adequate renal function: Calculated creatinine clearance >/= 30ml/min
* Be able to lie comfortably on back for 1 hour

Exclusion Criteria for Cancer Patients:

* As judged by investigator evidence of systemic disease that makes unsuitable for study
* Contra-indication for serial MRI scans
* Previous solid tumor treated within last 5 years
* Pregnancy
* History of significant obstructive airway disease
* History of gadolinium contrast allergy

Inclusion Criteria for Healthy Volunteers

* Age >/= 18 years
* Able to receive and understand verbal and written information regarding study and able to give written informed consent
* Willingness to undergo repeat MRI

Exclusion Criteria for Healthy Volunteers

* Unwillingness to sign informed consent
* Contra-indication for MRI
* Underlying significant respiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in hypoxia level during radiotherapy as assessed by fMRI (functional magnetic resonance imaging) | Baseline, Week 2 and 4 of radiotherapy, Week 6-8 post radiotherapy
  fMRI images will be used to assess tumour hypoxia status for Head and Neck Squamous Cell Carcinoma (HNSCC)
Change in tumour tissue and microenvironment during radiotherapy as assessed by fMRI | Weekly MRI imaging during radiotherapy (Up to 7 weeks)
  fMRI images will be used to evaluate on treatment tumour response to determine the effect of dose escalation to tumor sub regions using a daily online adaptive radiation treatment approach

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McPartlin, MD, Principal Investigator — Radiation Oncologist
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No